CLINICAL TRIAL: NCT05183997
Title: Effect of Verapamil as an Adjuvant to Bupivacaine in Supraclavicular Brachial Plexus Block Guided by Ultrasound for Forearm and Hand Surgeries
Brief Title: Verapamil in Supraclavicular Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hosny Sayed, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: vsbpb
Record Dates: First submitted 2021-10-08; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Regional Anesthesia Morbidity
MeSH Terms: interventions — Blood Cell Count; Prothrombin Time; Verapamil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) : 30 patients (control group): (Placebo Comparator): Patient will receive 20 to 30 ml bupivacaine plus 2 ml of normal saline .
  Interventions: Diagnostic Test: complete blood count; Diagnostic Test: prothrombin time; Diagnostic Test: prothrombin concentration
- Group (B) : 30 patients (verapamil group): (Experimental): Patient will receive 20 to 30 ml bupivacaine plus 5 mg of verapamil diluted in 2 ml of normal saline.
  Interventions: Diagnostic Test: complete blood count; Diagnostic Test: prothrombin time; Diagnostic Test: prothrombin concentration; Drug: Verapamil

INTERVENTIONS:
Diagnostic Test: complete blood count — laboratory test
Diagnostic Test: prothrombin time — laboratory test
Diagnostic Test: prothrombin concentration — laboratory test
Drug: Verapamil — drug will be add to prolong the effect of regional block
  Other Names: Isoptin
  Arms: Group (B) : 30 patients (verapamil group):

SUMMARY:
Supraclavicular brachial plexus block (SCBPB) is the common approach to provide surgical anesthesia of upper limb. The effects of single-injection brachial plexus nerve blocks recede after several hours unmasking the moderate to- severe pain of the surgical insult.

DETAILED DESCRIPTION:
Strategies to prolong brachial plexus nerve blocks analgesia beyond the pharmacological duration of the local anaesthetic used include placement of indwelling perineural catheters to allow prolonged infusion or the co-administration of adjuvants such as epinephrine, a2 agonists (i.e. clonidine and dexmedetomidine), midazolam, or the corticosteroid dexamethasone.

The investigators will use calcium channel blocker as adjuvant to bupivacaine in supraclavicular block. Calcium plays an important role in analgesia produced by local anesthetics. The activation of N-methyl-D-aspartate receptors may lead to calcium entry into cells and potentiation of spinal cord and plays a role in pain formation. Hence, calcium channel blockers may prevent central sensitization and provide better sensory motor block characteristics. Verapamil, a calcium channel blocker can potentiate analgesic action of local anesthetics and reduce postoperative pain and analgesic consumption. Few studies were there using 2.5 mg of verapamil, showing no effect on onset and duration of sensory motor block. Hence, the investigators have used 5 mg of verapamil as adjuvant to bupivacaine. The primary aim of the study was to know whether verapamil (5 mg) as adjuvant to bupivacaine in supraclavicular brachial plexus block would delay the need of rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients older than 18years and scheduled for forearm and hand surgeries like :

  1. fracture radius and ulna.
  2. cut wrists.

Exclusion Criteria:

1. allergy to the study drugs,
2. skin infection at site of needle puncture,
3. significant organ dysfunction, coagulopathy, drug or alcohol abuse, epilepsy, and psychiatric illness that would interfere with perception and assessment of pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
duration of postoperative analgesia. | in first 24 hours
  blinded observer will collect the Visual Analogue Score (VAS) for pain scored from Zero to ten where 0= no pain and 10 = the worst pain imaginable for acute post-operative pain.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Knezevic NN, Anantamongkol U, Candido KD. Perineural dexamethasone added to local anesthesia for brachial plexus block improves pain but delays block onset and motor blockade recovery. Pain Physician. 2015 Jan-Feb;18(1):1-14. PMID 25675053
- [Background] Popping DM, Elia N, Marret E, Wenk M, Tramer MR. Clonidine as an adjuvant to local anesthetics for peripheral nerve and plexus blocks: a meta-analysis of randomized trials. Anesthesiology. 2009 Aug;111(2):406-15. doi: 10.1097/ALN.0b013e3181aae897. PMID 19602964
- [Background] Malmberg AB, Yaksh TL. Voltage-sensitive calcium channels in spinal nociceptive processing: blockade of N- and P-type channels inhibits formalin-induced nociception. J Neurosci. 1994 Aug;14(8):4882-90. doi: 10.1523/JNEUROSCI.14-08-04882.1994. PMID 8046458
- [Background] Brose WG, Gutlove DP, Luther RR, Bowersox SS, McGuire D. Use of intrathecal SNX-111, a novel, N-type, voltage-sensitive, calcium channel blocker, in the management of intractable brachial plexus avulsion pain. Clin J Pain. 1997 Sep;13(3):256-9. doi: 10.1097/00002508-199709000-00012. PMID 9303259